CLINICAL TRIAL: NCT00704015
Title: Smoking Cessation Intervention in Acute Orthopedic Surgery - A Randomized Controlled Trial
Brief Title: Smoking Cessation Intervention in Acute Orthopedic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Sari Ponzer. MD, Prof, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 03-215
Record Dates: First submitted 2008-06-23; First posted 2008-06-24 (Estimated); Last update posted 2008-06-24 (Estimated); Status verified 2008-06

CONDITIONS: Smoking Cessation; Fracture
Keywords: Smoking cessation; Acute injury; Musculoskeletal; Postoperative complications
MeSH Terms: conditions — Smoking Cessation; Fractures, Bone; Postoperative Complications

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Smoking cessation
  Interventions: Behavioral: Smoking cessation
- B (No Intervention)

INTERVENTIONS:
Behavioral: Smoking cessation — Nurses, specifically trained for smoking cession program, contacted the patients at the orthopedic wards and initiated the intervention (stop smoking) within 1-2 days after acute hospitalization. The intervention included one or two personal meetings and weekly phone contacts during 6 weeks with a trained nurse. A phone number to a non-smoking hotline was provided for all patients. The patients were continuously encouraged not to smoke and free nicotine substitution (Nicorette®) was offered those who needed it. No other drug therapy was used.
  Arms: A

SUMMARY:
The purpose of this study was to evaluate if an intervention with smoking cessation starting during the acute hospitalization period and continuing during the acute postoperative phase of 6 weeks would reduce the frequency of overall postoperative complications and wound infections in patients with acute musculoskeletal injuries requiring surgical treatment. The secondary aims were to study the short and the long term (1 year) abstinence rate, functional outcome, health related quality of life as well as costs.

DETAILED DESCRIPTION:
Tobacco smoking is a major health problem. The effect of a smoking cessation intervention prior to elective orthopedic surgery has been evaluated previously. However, as far as we know there are no prospective randomized studies investigating the effect of smoking cessation on complication rate in patients with acute musculoskeletal injuries.

ELIGIBILITY:
Inclusion Criteria:

* daily smoker: more than 2 cigarettes per day for at least one year
* acute fracture of an extremity, in need of surgical treatment
* oral and written consent

Exclusion Criteria:

* pregnancy
* alcohol or drug abuse prohibiting compliance with the study protocol
* living outside the county of Stockholm prohibiting follow-up
* a severe mental illness including dementia
* inability to read and understand Swedish

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2004-02; Primary Completion 2006-12 (Actual); Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications including wound related complications | 6-12 weeks

SECONDARY OUTCOMES:
Abstinence rate and functional outcome including HRQoL | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sari Ponzer, MD, Prof, Principal Investigator — Karolinska Institutet